CLINICAL TRIAL: NCT00663871
Title: BioBehavioral Studies of Cardiovascular Disease
Brief Title: Evaluating the Effects of Omega-3 Fatty Acids on Heart Disease and Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Stephen Manuck, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY19060029; 2P01HL040962 (NIH); R01AT004699 (NIH)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2021-05-12 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Diseases; Mood Disorders; Inflammation
Keywords: Fish Oil; Omega-3 fatty acids; Affect; Depression; Anger; Nutrition; Impulsivity; Aggression; Cognition; Behavior
MeSH Terms: conditions — Cardiovascular Diseases; Mood Disorders; Inflammation; Depression; Impulsive Behavior; Aggression; Behavior | interventions — Fish Oils; Soybean Oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish Oil (Active Comparator): Participants will take fish oil supplements daily for 4 months.
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): Participants will take soybean oil (placebo) supplements daily for 4 months.
  Interventions: Dietary Supplement: Soybean Oil (Placebo)

INTERVENTIONS:
Dietary Supplement: Fish Oil — Participants will take 2 grams (1400 mg EPA and DHA) of fish oil supplements on a daily basis.
  Other Names: Omega-3 Life Formula (PharmaOmega)
  Arms: Fish Oil
Dietary Supplement: Soybean Oil (Placebo) — Participants will take 2 grams of soybean oil supplements on a daily basis.
  Arms: Placebo

SUMMARY:
Omega-3 fatty acids are a certain kind of fish fat that has recently been shown to have health benefits. This study will examine the effectiveness of fish oil supplementation for reducing the early signs of heart disease risk and for improving mood, impulsivity, and anger levels.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a broad term that includes diseases that affect the heart and blood vessels, including coronary heart disease, heart failure, high blood pressure, stroke and vascular dementia. CVD is the leading cause of death in the United States, resulting in 700,000 deaths each year. Preliminary research has shown that increased consumption of fish, specifically the omega-3 fatty acids found in fish oil, has beneficial effects in people with CVD. Fish oil may also have positive effects on the psychological health and well-being of people with psychiatric disorders. However, more research is needed to confirm the positive physical and psychological effects of fish oil in healthy adults. The purpose of this study is to explore potentail effects of fish oil supplementation on CVD mechanisms and risk markers, and on depressive symptoms, antagonistic disposition, and levels of impulsivity and aggression.

This study will enroll healthy adults who habitually consume low quantities of long-chain omega-3 fatty acids. Participants will be randomly assigned to receive either fish oil supplements or placebo on a daily basis for 4 months. Study visits will occur at baseline and Months 2 and 4. At the baseline and Month 4 visits, participants will undergo the following measures as primary study aims: blood collection for inflammatory markers; heart rate and variability measurements; and interviews, psychological tests, and questionnaires to assess mood, disposition, impulsivity, and aggression.

As secondary aims, we will test for any effects of fish oil on cognitive performance and, if a main effect on inflammatory markers is found, we will test for moderation by select genetic polymorphisms.

As an exploratory aim, we will test for any effects of fish oil on structural or functional brain imaging. (This exploratory aim was mistakenly listed as a secondary aim at the time of trial registration.)

ELIGIBILITY:
Inclusion Criteria:

* Currently employed at least 25 hours a week, but does not regularly work the third shift (i.e., night shift)
* English is primary language
* Consumes less than 300 mg/day of long-chain omega-3 fatty acids.

Exclusion Criteria:

* Serious allergy to fish (e.g., anaphylaxis, bronchospasm, serious skin reaction)
* History of atherosclerotic disease (e.g., myocardial infarction) or treatment of angina or claudication (e.g., angioplasty)
* Reported history of schizophrenia or bipolar disorder
* Long-term hepatitis
* Kidney failure
* Stroke or other neurological disorder
* Lung disease requiring drug treatment
* Stage 2 high blood pressure, defined as systolic blood pressure of 160 mm Hg or greater and diastolic blood pressure of 100 mm Hg or greater
* Alcohol consumption of more than five drinks per day each week (i.e., more than 35 alcoholic drinks each week)
* Pregnant or breastfeeding
* Currently taking any cardiovascular, psychotropic, glucocorticoid, lipid-lowering, insulin, or weight loss medications
* Currently taking fish oil supplements

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 272 (Actual)
Dates: Start 2008-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew F. Muldoon, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muldoon MF, Ryan CM, Yao JK, Conklin SM, Manuck SB. Long-chain omega-3 fatty acids and optimization of cognitive performance. Mil Med. 2014 Nov;179(11 Suppl):95-105. doi: 10.7205/MILMED-D-14-00168. PMID 25373092
- [Result] Leckie RL, Lehman DE, Gianaros PJ, Erickson KI, Sereika SM, Kuan DCH, Manuck SB, Ryan CM, Yao JK, Muldoon MF. The effects of omega-3 fatty acids on neuropsychological functioning and brain morphology in mid-life adults: a randomized clinical trial. Psychol Med. 2020 Oct;50(14):2425-2434. doi: 10.1017/S0033291719002617. Epub 2019 Oct 4. PMID 31581959
- [Result] Muldoon MF, Laderian B, Kuan DC, Sereika SM, Marsland AL, Manuck SB. Fish oil supplementation does not lower C-reactive protein or interleukin-6 levels in healthy adults. J Intern Med. 2016 Jan;279(1):98-109. doi: 10.1111/joim.12442. Epub 2015 Oct 26. PMID 26497831
- [Result] Ginty AT, Muldoon MF, Kuan DCH, Schirda B, Kamarck TW, Jennings JR, Manuck SB, Gianaros PJ. Omega-3 Supplementation and the Neural Correlates of Negative Affect and Impulsivity: A Double-Blind, Randomized, Placebo-Controlled Trial in Midlife Adults. Psychosom Med. 2017 Jun;79(5):549-556. doi: 10.1097/PSY.0000000000000453. PMID 28121722
- [Result] Cipollina C, Salvatore SR, Muldoon MF, Freeman BA, Schopfer FJ. Generation and dietary modulation of anti-inflammatory electrophilic omega-3 fatty acid derivatives. PLoS One. 2014 Apr 15;9(4):e94836. doi: 10.1371/journal.pone.0094836. eCollection 2014. PMID 24736647
- [Result] Muldoon MF, Ryan CM, Sheu L, Yao JK, Conklin SM, Manuck SB. Serum phospholipid docosahexaenonic acid is associated with cognitive functioning during middle adulthood. J Nutr. 2010 Apr;140(4):848-53. doi: 10.3945/jn.109.119578. Epub 2010 Feb 24. PMID 20181791
- [Result] Liu JC, Conklin SM, Manuck SB, Yao JK, Muldoon MF. Long-chain omega-3 fatty acids and blood pressure. Am J Hypertens. 2011 Oct;24(10):1121-6. doi: 10.1038/ajh.2011.120. Epub 2011 Jul 14. PMID 21753804
- [Result] Conklin SM, Harris JI, Manuck SB, Yao JK, Hibbeln JR, Muldoon MF. Serum omega-3 fatty acids are associated with variation in mood, personality and behavior in hypercholesterolemic community volunteers. Psychiatry Res. 2007 Jul 30;152(1):1-10. doi: 10.1016/j.psychres.2006.10.006. Epub 2007 Mar 23. PMID 17383013
- [Result] Conklin SM, Gianaros PJ, Brown SM, Yao JK, Hariri AR, Manuck SB, Muldoon MF. Long-chain omega-3 fatty acid intake is associated positively with corticolimbic gray matter volume in healthy adults. Neurosci Lett. 2007 Jun 29;421(3):209-12. doi: 10.1016/j.neulet.2007.04.086. Epub 2007 Jun 2. PMID 17574755
- [Result] Conklin SM, Manuck SB, Yao JK, Flory JD, Hibbeln JR, Muldoon MF. High omega-6 and low omega-3 fatty acids are associated with depressive symptoms and neuroticism. Psychosom Med. 2007 Dec;69(9):932-4. doi: 10.1097/PSY.0b013e31815aaa42. Epub 2007 Nov 8. PMID 17991818
- [Result] Conklin SM, Runyan CA, Leonard S, Reddy RD, Muldoon MF, Yao JK. Age-related changes of n-3 and n-6 polyunsaturated fatty acids in the anterior cingulate cortex of individuals with major depressive disorder. Prostaglandins Leukot Essent Fatty Acids. 2010 Feb-Mar;82(2-3):111-9. doi: 10.1016/j.plefa.2009.12.002. Epub 2010 Jan 8. PMID 20060277
- [Result] Muldoon MF, Erickson KI, Goodpaster BH, Jakicic JM, Conklin SM, Sekikawa A, Yao JK, Manuck SB. Concurrent physical activity modifies the association between n3 long-chain fatty acids and cardiometabolic risk in midlife adults. J Nutr. 2013 Sep;143(9):1414-20. doi: 10.3945/jn.113.174078. Epub 2013 Jul 24. PMID 23884386

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fish Oil | Placebo
Started | 134 | 138
Completed | 124 | 131
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil | Placebo | Total
Number analyzed (Participants) | 134 | 138 | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 134 | 138 | 272
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 78 | 154
  Male | 58 | 60 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 132 | 136 | 268
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 22 | 43
  White | 109 | 116 | 225
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 134 | 138 | 272

OUTCOME MEASURES:

1. Primary Outcome: Circulating Serum Interleukin-6 (IL-6)
Description: Systemic inflammation: fasting serum Interleukin-6 (IL-6)
Time Frame: Baseline and Month 4
Population: 11 participants had chronic inflammatory conditions at baseline and were excluded, leaving 129 in fish oil and 132 in placebo groups.
  The 17 subjects who did not finish the study were retained through use of single-imputation analysis. Any subject missing both baseline and 4-month data could not be retained. TThis applied to 2 fish oil and 1 placebo participants for IL-6, leaving 127 and 131, respectively in the analysis population.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 127 | 131
pg/mL
  baseline | 1.13 [0.465 to 1.79] | 1.01 [0.60 to 1.40]
  Month 4 | 0.88 [0.60 to 1.72] | 0.81 [0.53 to 1.31]
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.59, ANOVA; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.27 to 0.19]

2. Primary Outcome: C-reactive Protein (CRP)
Description: fasting serum C-reactive protein (CRP) in milligrams per liter (mg/L)
Time Frame: baseline and month 4
Population: 11 participants had chronic inflammatory conditions at baseline and were excluded, leaving 129 in fish oil and 132 in placebo groups.
  The 17 subjects who did not finish the study were retained through use of single-imputation analysis. Any subject missing both baseline and 4-month data could not be retained. This applied to 4 fish oil and 3 placebo participants for CRP, leaving 125 and 129, respectively, in the analysis population.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 125 | 129
mg/L
  baseline | 1.00 [.043 to 2.17] | 0.67 [0.30 to 1.67]
  month 4 | 0.94 [.042 to 2.02] | 0.64 [0.33 to 1.87]
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.21, ANOVA; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.24 to 0.19]

3. Primary Outcome: Negative Affect
Description: Negative affect questions adapted from the Positive and Negative Affect Schedule - Expanded Form administered via ecological momentary assessment. The minimum value is 1, and the maximum value is 6. A higher score are worse (more negative affect).
Time Frame: baseline and month 4
Population: All randomized participants were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 138
units on a scale
  Baseline | 1.76 [1.23 to 2.42] | 1.69 [1.28 to 2.45]
  Month 4 | 1.73 [1.20 to 2.33] | 1.59 [1.21 to 2.34]
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.92, Mixed Models Analysis — The model included effects of treatment (fish oil, placebo), time (baseline, post-intervention), and interaction terms of treatment with time. The Negative Affect scores were categorized by quartiles of the baseline measures; Generalized Linear Mixed Modeling was used with a multinomial distribution with cumulative link; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.69 to 1.50]

4. Primary Outcome: Impulsivity
Description: Barratt Impulsiveness Scale. The minimum value is 34, and the maximum value is 120. A higher score suggests a worse outcome.
Time Frame: baseline and month 4
Population: All randomized participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 138
units on a scale
  Baseline | 60.44 (8.53) | 59.57 (8.44)
  Month 4 | 60.41 (9.27) | 59.38 (8.97)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.86, Mixed Models Analysis — The model included effects of treatment (fish oil, placebo), time (baseline, post-intervention), and interaction terms of treatment with time; Mean Difference (Net) = 0.12, 95% CI 2-sided [-1.21 to 1.44]

5. Primary Outcome: Aggression
Description: Bus-Perry Aggression Questionnaire. The minimum value is 14, and the maximum value is 53. A higher score suggests a worse outcome.
Time Frame: baseline and month 4
Population: All randomized participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 138
units on a scale
  Baseline | 28.14 (8.32) | 27.55 (7.51)
  Month 4 | 27.75 (8.90) | 27.46 (7.72)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.63, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = -0.31, 95% CI 2-sided [-1.57 to 0.94]

6. Primary Outcome: Hostility, Barefoot Score
Description: The 27-item Barefoot Hostility Scale. The minimum value is 1, and the maximum value is 30. A higher score suggests a worse outcome.
Time Frame: baseline and month 4
Population: All randomized participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 138
units on a scale
  Baseline | 13.58 (6.52) | 12.54 (6.21)
  Month 4 | 13.30 (6.53) | 12.58 (6.13)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.50, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = -0.32, 95% CI 2-sided [-1.25 to 0.61]

7. Primary Outcome: Trait Anger
Description: State-Trait Anger Expression Inventory. The minimum value is 10, and the maximum value is 40. A higher score suggests a worse outcome.
Time Frame: baseline and month 4
Population: All randomized participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 138
units on a scale
  Baseline | 16.07 (3.69) | 16.01 (3.33)
  Month 4 | 15.39 (3.32) | 15.03 (3.21)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.25, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = 0.33, 95% CI 2-sided [-0.23 to 0.88]

8. Primary Outcome: Anger Expression
Description: State-Trait Anger Expression Inventory. The minimum value is 0, and the maximum value is 72. A higher score suggests a worse outcome.
Time Frame: baseline and month 4
Population: All randomized participants were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 138
units on a scale
  Baseline | 24.73 (8.86) | 24.50 (8.38)
  Month 4 | 22.83 (8.63) | 23.25 (7.77)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.52, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Net) = -0.45, 95% CI 2-sided [-1.83 to 0.92]

9. Primary Outcome: Type A, Total Score
Description: Structured Interview - Type A Behavior Pattern using the Interpersonal Hostility Assessment Technique (IHAT). The minimum value is 0, and the maximum value is 12. A higher score suggests a worse outcome.
Time Frame: baseline and month 4
Population: All randomized participants were analyzed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 138
units on a scale
  Baseline | 1.0 [0 to 2.5] | 1.0 [0 to 2.0]
  Month 4 | 1.0 [0 to 2.0] | 1.0 [0.5 to 1.83]
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.52, Mixed Models Analysis — The model included effects for treatment (fish oil, placebo), time (baseline, post-intervention), and interaction terms of treatment with time. The Type A personality scores were categorized by quartiles of the baseline measures; Generalized Linear Mixed Modeling was used with a multinomial distribution with cumulative link; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.67 to 2.24]

10. Primary Outcome: Mean Successive Difference in Inter-beat Intervals Natural Log Transformed Paced Respiration
Description: Mean successive difference in inter-beat intervals natural log transformed paced respiration in milliseconds
Time Frame: baseline and month 4
Population: One participant was excluded from the analysis due to missing both at baseline and 4-month data..
Measure: Mean (Standard Deviation); unit: ln(milliseconds)
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
ln(milliseconds)
  Baseline | 2.99 (0.77) | 3.13 (0.69)
  Month 4 | 2.92 (0.83) | 3.08 (0.63)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.68, Mixed Models Analysis — The model included effects for treatment (fish oil, placebo), time (baseline, post-intervention), and interaction terms of treatment with time; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.16 to 0.10]

11. Primary Outcome: High Frequency (.12 to .40 Hz) Heart Rate Variability Natural Log Transformed Paced Respiration
Description: High frequency (.12 to .40 Hz) heart rate variability natural log transformed paced respiration in Hertz units (Hz)
Time Frame: baseline and month 4
Population: One participant was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: ln(hertz)
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
ln(hertz)
  Baseline | 5.93 (1.52) | 6.15 (1.38)
  Month 4 | 5.74 (1.66) | 6.13 (1.28)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other — The model included effects for treatment (fish oil, placebo), time (baseline, post-intervention), and interaction terms of treatment with time; p = 0.16, Mixed Models Analysis; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.41 to 0.07]

12. Primary Outcome: Total Power (0 to .40 Hz) Heart Rate Variability Natural Log Transformed Paced Respiration
Description: Total power (0 to .40 Hz) heart rate variability natural log transformed paced respiration in Hertz (Hz) units.
Time Frame: baseline and month 4
Population: One participant was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: ln(hertz)
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
ln(hertz)
  Baseline | 7.02 (1.10) | 7.21 (0.97)
  Month 4 | 6.94 (1.10) | 7.18 (0.92)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other — [test comment as in outcome 11, analysis 1]; p = 0.59, Mixed Models Analysis; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.24 to 0.14]

13. Primary Outcome: Mean Successive Difference in Inter-beat Intervals Natural Log Transformed Unpaced Respiration
Description: Mean successive difference in inter-beat intervals natural log transformed unpaced respiration in milliseconds (msec)
Time Frame: baseline and month 4
Population: One participant was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: ln(milliseconds)
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
ln(milliseconds)
  Baseline | 2.97 (0.71) | 3.11 (0.67)
  Month 4 | 2.95 (0.71) | 3.03 (0.59)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other — [test comment as in outcome 11, analysis 1]; p = 0.35, Mixed Models Analysis; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.06 to 0.18]

14. Primary Outcome: High Frequency (.12 to .40 Hz) Heart Rate Variability Natural Log Transformed Unpaced Respiration
Description: High frequency (.12 to .40 Hz) heart rate variability natural log transformed unpaced respiration in Hertz (Hz) units
Time Frame: baseline and month 4
Population: One participant was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: ln(hertz)
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
ln(hertz)
  Baseline | 5.37 (1.40) | 5.61 (1.28)
  Month 4 | 5.29 (1.41) | 5.51 (1.21)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other — [test comment as in outcome 11, analysis 1]; p = 0.74, Mixed Models Analysis; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.18 to 0.25]

15. Primary Outcome: Total Power (0 to .40 Hz) Heart Rate Variability Natural Log Transformed Unpaced Respiration
Description: Total power (0 to .40 Hz) heart rate variability natural log transformed unpaced respiration in Hertz (Hz) units
Time Frame: baseline and month 4
Population: One participant in placebo group was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: ln(hertz)
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
ln(hertz)
  Baseline | 7.05 (0.98) | 7.13 (0.97)
  Month 4 | 6.98 (0.97) | 7.15 (0.87)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other — [test comment as in outcome 11, analysis 1]; p = 0.28, Mixed Models Analysis; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.27 to 0.08]

16. Secondary Outcome: Executive Function
Description: Executive function was comprised of trail making B - A time, digit span forward and digit span backward completions. Performance scores on each task were converted into Z-scores, and then averaged across tasks. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate higher function (better outcome). The analysis compared changes in Z-scores between the two treatment groups.
Time Frame: Baseline and Month 4
Population: One participant in placebo group was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
Z-score
  baseline | -0.02 (0.57) | 0.02 (0.61)
  Month 4 | 0.07 (0.62) | 0.03 (0.63)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.76, Repeated Measures MANOVA; standardized mean difference = 0.15, 95% CI 2-sided [-0.09 to 0.39]

17. Secondary Outcome: Learning / Episodic Memory
Description: Learning/episodic memory was comprised of d' from the four word memory task and the average performance across all trials of the Rey auditory verbal learning test. Performance scores on each task were converted into Z-scores, and then averaged across tasks. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate higher function (better outcome). The analysis compared changes in Z-scores between the two treatment groups.
Time Frame: Baseline and Month 4
Population: One participant in placebo group was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
Z-score
  baseline | 0.01 (0.87) | -0.01 (0.86)
  Month 4 | 0.18 (0.85) | 0.12 (0.87)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.62, Repeated Measures MANOVA; standardized mean difference = 0.06, 95% CI 2-sided [-0.18 to 0.30]

18. Secondary Outcome: Psychomotor Speed
Description: Psychomotor speed was comprised of trail making A time, Stroop word-only time and color-only time. Performance scores on each task were converted into Z-scores, and then averaged across tasks. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate higher function (better outcome). The analysis compared changes in Z-scores between the two treatment groups.
Time Frame: Baseline and Month 4
Population: One participant in placebo group was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
Z-score
  baseline | 0.04 (0.63) | -0.04 (0.60)
  Month 4 | 0.13 (0.54) | 0.007 (0.57)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.42, Repeated Measures MANOVA; standardized mean difference = 0.03, 95% CI 2-sided [-0.21 to 0.26]

19. Secondary Outcome: Fluid Intelligence
Description: This outcome was based upon matrix reasoning task raw score, block design task raw score and spatial span forward raw score. Performance scores on each task were converted into Z-scores, and then averaged across tasks. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z scores indicate higher function (better outcome). The analysis compared changes in Z-scores between the two treatment groups.
Time Frame: Baseline and Month 4
Population: One participant in placebo group was excluded from the analysis due to missing both at baseline and 4-month data.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 134 | 137
Z-score
  baseline | -0.02 (0.85) | 0.02 (0.90)
  Month 4 | -0.005 (0.82) | 0.05 (0.83)
Statistical Analysis 1: Comparison: Fish Oil vs Placebo; Test type: Superiority or Other; p = 0.54, Repeated Measures MANOVA; Repeated Measures MANOVA; Standardized mean difference = -0.06, 95% CI 2-sided [-0.30 to 0.18]

20. Secondary Outcome: Moderation of Effects of Fish Oil on Inflammatory Markers by Select Genetic Polymorphisms
Description: Circulating serum concentrations of IL6 and CRP before and after supplementation with fish oil or placebo.
Time Frame: Measured at Month 4
Population: This aim was conditional and was not completed per the protocol.
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 0 | 0

21. Other Pre Specified Outcome: Structural & Functional MRI
Description: Measures of brain structure and function from magnetic resonance imaging
Time Frame: Baseline and month 4
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 months
Description: Used pre-specified 9 item side effect questionnaire.
Arm/Group | Fish Oil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/134 | 0/138
Other Adverse Events (participants affected / at risk) | 61/134 | 17/138
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil (N=134) | Placebo (N=138)
Fishy belch or after-taste (General disorders) | 51 (51) | 14 (14)
Loose stool, bloating or gas pains (Gastrointestinal disorders) | 10 (10) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No